CLINICAL TRIAL: NCT04789148
Title: Effects of Intranasal Oxytocin in Patients With Arginine-vasopressin Deficiency - A Pilot Study
Brief Title: Effects of Intranasal Oxytocin in Patients With Arginine-vasopressin Deficiency
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Elizabeth Austen Lawson (Other)
Collaborators: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Austen Lawson, Associate Professor of Medicine, Harvard Medical School; Director, Interdisciplinary Oxytocin Research Program, Neuroendocrine Unit, Massachusetts General Hospital, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020P003071
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Vasopressin Deficiency
Keywords: Hypopituitarism; posterior pituitary; oxytocin; psychopathology; anxiety; depressive symptoms; socioemotional functioning
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Hypopituitarism; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, single dose crossover study evaluating 2 different dose levels of intranasal oxytocin vs placebo (Part A), followed by Part B, an optional 2-week randomized, double-blind, placebo-controlled substudy investigating intranasal oxytocin 6 IU vs. placebo three times a day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A Arm 1 (Experimental): Main visit 1: 6 IU intranasal oxytocin; Main visit 2: 24 IU intranasal oxytocin; Main visit 3: intranasal placebo
  Interventions: Drug: Intranasal Oxytocin (IN-OXT); Drug: Placebo
- Part A Arm 2 (Experimental): Main visit 1: 6 IU intranasal oxytocin; Main visit 2: intranasal placebo; Main visit 3: 24 IU intranasal oxytocin
  Interventions: Drug: Intranasal Oxytocin (IN-OXT); Drug: Placebo
- Part A Arm 3 (Experimental): Main visit 1: 24 IU intranasal oxytocin; Main visit 2: 6 IU intranasal oxytocin; Main visit 3: intranasal placebo
  Interventions: Drug: Intranasal Oxytocin (IN-OXT); Drug: Placebo
- Part A Arm 4 (Experimental): Main visit 1: 24 IU intranasal oxytocin; Main visit 2: intranasal placebo; Main visit 3: 6 IU intranasal oxytocin
  Interventions: Drug: Intranasal Oxytocin (IN-OXT); Drug: Placebo
- Part A Arm 5 (Experimental): Main visit 1: intranasal placebo; Main visit 2: 6 IU intranasal oxytocin; Main visit 3: 24 IU intranasal oxytocin
  Interventions: Drug: Intranasal Oxytocin (IN-OXT); Drug: Placebo
- Part A Arm 6 (Experimental): Main visit 1: intranasal placebo; Main visit 2: 24 IU intranasal oxytocin; Main visit 3: 6 IU intranasal oxytocin
  Interventions: Drug: Intranasal Oxytocin (IN-OXT); Drug: Placebo
- Part B Arm 1 (Active Comparator): Intranasal oxytocin 6 IU three times a day for 14 days
  Interventions: Drug: Intranasal Oxytocin (IN-OXT)
- Part B Arm 2 (Experimental): Intranasal placebo three times a day for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin (IN-OXT) — 6 IU single dose
  Arms: Part A Arm 1; Part A Arm 2; Part A Arm 3; Part A Arm 4; Part A Arm 5; Part A Arm 6
Drug: Intranasal Oxytocin (IN-OXT) — IN-OXT 6 IU three times a day for 2 weeks
  Arms: Part A Arm 1; Part A Arm 2; Part A Arm 3; Part A Arm 4; Part A Arm 5; Part A Arm 6
Drug: Placebo — Intranasal placebo three times a day for 2 weeks
  Arms: Part A Arm 1; Part A Arm 2; Part A Arm 3; Part A Arm 4; Part A Arm 5; Part A Arm 6
Drug: Intranasal Oxytocin (IN-OXT) — 24 IU single dose
  Arms: Part B Arm 1
Drug: Placebo — placebo single dose
  Arms: Part B Arm 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled crossover pilot study of single-dose intranasal oxytocin (6 IU and 24 IU) vs. placebo in adult men and women (aged 18 years and above) with arginine-vasopressin deficiency to evaluate the effect of oxytocin on anxiety, depression, and socioemotional functioning (Part A), with an optional randomized, double-blind, placebo-controlled 2-week repeated dose substudy of intranasal oxytocin 6 IU or placebo (Part B).

Following a screening visit to determine eligibility, participants will return for three main study visits in Part A. During the main study visits, study participants will receive either oxytocin or placebo, followed by assessments of emotional behavior.

In Part A, thirty participants will be equally randomized to one of six possible groups:

1. 6 IU oxytocin - 24 IU oxytocin - placebo
2. 6 IU oxytocin - placebo - 24 IU oxytocin
3. 24 IU oxytocin - 6 IU oxytocin - placebo
4. 24 IU oxytocin - placebo - 6 IU oxytocin
5. placebo - 6 IU oxytocin - 24 IU oxytocin
6. placebo - 24 IU oxytocin - 6 IU oxytocin

Following completion of the Part A crossover portion of the study, in Part B participants may also choose to continue participation in an optional, randomized, double-blind, placebo-controlled substudy of intranasal oxytocin 6 IU or placebo three times a day for two weeks, followed by assessments of emotional behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Arginine-vasopressin deficiency
* Normal FT4 or T4
* Normal serum/plasma sodium
* Stable hormone replacement

Exclusion Criteria:

* Active substance use disorder within the last 6 months
* History of psychosis
* Suicidal behavior and/or active suicidal ideation with plan and/or intent, e.g., suicidal ideation of type 4 or type 5 as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS), in the last month
* Medication changes within 4 weeks of enrollment or planned medication changes during the study
* History of chronic nasal obstruction or local pathology in nostril pathway which, in the opinion of the investigator, would prevent appropriate nasal administration of the study drug.
* History of cardiac disease, including arrhythmias, coronary heart disease, coronary artery spasms, valvular heart disease, hypertrophic cardiomyopathy (hypertension is not exclusionary)
* History of chronic kidney disease stage III and above
* History of liver cirrhosis
* Pregnancy or breastfeeding within the last 8 weeks
* Unwilling to use a medically acceptable form of contraception throughout the study period (female of child-bearing potential only)
* Any significant illness, condition, drug or medical device that the Investigator determines could interfere with study participation, data collection, or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dot-probe task - anxious behavior between low dose oxytocin and placebo | 20 minutes following intervention at each main visit
  Difference in response times (in milliseconds) to dots appearing in the location of the previously shown negative versus the neutral face between 6 IU oxytocin vs placebo in the dot-probe task.

SECONDARY OUTCOMES:
Dot-probe task - anxious behavior between all three interventions | 20 minutes following intervention
  Difference in response time (in milliseconds) to dots appearing in the location of the previously shown negative versus neutral face between 6 IU oxytocin, 24 IU oxytocin, and placebo in the dot-probe task.
Depressive behavior - probabilistic reward task between all three interventions | 30 minutes following intervention at each main visit
  Response bias developed toward the more frequently reinforced alternative between 6 IU oxytocin, 24 IU oxytocin, and placebo in the probabilistic reward task.
Socioemotional functioning - Emotion recognition task between all three interventions | 40 minutes following intervention at each main visit
  Accuracy in identifying correct emotion between 6 IU oxytocin, 24 IU oxytocin, and placebo in the emotion recognition task.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Neuroendocrine Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No